CLINICAL TRIAL: NCT03624465
Title: Prospective Clinical Study of the Levita Magnetics Surgical System Used for Prostatectomy Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Levita Magnetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CP005
Record Dates: First submitted 2018-08-07; First posted 2018-08-10 (Actual); Results first posted 2024-12-12 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Prostatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Levita Magnetic Surgical System (Experimental): Levita Magnetic Surgical System use of surgical tool
  Interventions: Device: Levita Magnetic Surgical System

INTERVENTIONS:
Device: Levita Magnetic Surgical System — Device for use as a surgical tool.

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the Levita Magnetic Surgical System in patients undergoing prostatectomy surgery.

DETAILED DESCRIPTION:
Prospective, multicenter, single-arm, open label study designed to assess the safety and effectiveness of the Levita Magnetic Surgical System in prostatectomy surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age
* Subject is scheduled to undergo elective prostatectomy surgery

Exclusion Criteria:

* Significant comorbidities
* Subjects with pacemakers, defibrillators, or other electromedical implants
* Subjects with ferromagnetic implants
* Clinical history of impaired coagulation
* Subject has an anatomical abnormality noted after initiation of index procedure that would prevent device use
* Subject is not likely to comply with the follow-up evaluation schedule
* Subject is participating in another clinical trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Gettman, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Fundacion Arturo Lopez Perez (FALP), Santiago, Chile

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Levita Magnetic Surgical System
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Levita Magnetic Surgical System
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Chile | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Tools Required to Retract the Prostate During Procedure
Description: Ability to adequately retract the prostate to achieve an effective exposure of the target tissue. Adequate retraction is achieved if it is not necessary to replace the Levita Magnetic Surgical System with another instrument to retract the prostate during the procedure.
Time Frame: During planned prostatectomy procudure
Measure: Number; unit: Additional Tools to Mobilize Liver
Arm/Group | Levita Magnetic Surgical System
Number analyzed (Participants) | 30
Additional Tools to Mobilize Liver | 0

2. Primary Outcome: Incidence of Device Related Adverse Events (Safety)
Description: All adverse events will be recorded and allocated as to relatedness to device, procedure or other.
Time Frame: Through 30 days post prostatectomy procedure.
Measure: Number; unit: Device Related AEs
Arm/Group | Levita Magnetic Surgical System
Number analyzed (Participants) | 30
Device Related AEs | 0

ADVERSE EVENTS:
Time Frame: Through 30 days post procedure.
Description: All adverse events were recorded and allocated as to relatedness to device, procedure, or other.
Arm/Group | Levita Magnetic Surgical System
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 10/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levita Magnetic Surgical System (N=30)
Minor bleeding from surgical site on left flank (Surgical and medical procedures) | 1 (1)
Ecchymosis in Assistant Port (Surgical and medical procedures) | 3 (3)
Chest Pain (General disorders) | 1 (1) — Investigator further detailed: "lasting for 30 min. (ECG, CK, CKMB and troponin "normal"
Meatal Stenosis (General disorders) | 1 (1)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal Wall Hematoma in Assistant Port Placement (Surgical and medical procedures) | 2 (2)
Ecchymosis Around Surgical Sites and Base of Penis Scrotum (Surgical and medical procedures) | 1 (1)
Infected Pelvic Lymphoceles (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/65/NCT03624465/Prot_SAP_000.pdf